CLINICAL TRIAL: NCT00371293
Title: Inflammatory Response to Sleep Apnea in Obese Subjects: The Cardiovascular Effects of Obstructive Sleep Apnea (COSA) Study
Brief Title: The Effects of Obesity and Obstructive Sleep Apnea on Inflammation and Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Julio A. Chirinos, MD, PhD, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 442; R01HL080076-01A1 (NIH)
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Sleep Apnea Syndromes; Inflammation
Keywords: Sleep Apnea; C-Reactive Protein; Obesity; Insulin Resistance; Arterial stiffness
MeSH Terms: conditions — Sleep Apnea Syndromes; Inflammation; Obesity; Insulin Resistance | interventions — Weight Reduction Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Participants will receive CPAP therapy.
  Interventions: Device: CPAP therapy
- 2 (Active Comparator): Participants will take part in a weight loss program.
  Interventions: Behavioral: Weight Loss Program
- 3 (Experimental): Participants will receive CPAP therapy and take part in a weight loss program.
  Interventions: Behavioral: Weight Loss Program; Device: CPAP therapy

INTERVENTIONS:
Behavioral: Weight Loss Program — Participants in the weight loss program will receive weekly dietary counseling and will be encouraged to decrease caloric intake and increase physical activity.
  Arms: 2; 3
Device: CPAP therapy — Participants receiving CPAP therapy will use a CPAP machine each night while they sleep.
  Arms: 1; 3

SUMMARY:
Obstructive sleep apnea (OSA) is a serious sleep disorder in which a person's breathing is restricted during sleep. Obese individuals with OSA are at an increased risk of inflammation and heart conditions, but it is unknown whether this risk is related to the effects of OSA or obesity. This study will evaluate whether OSA or obesity plays the primary role in inflammation related to heart disease. The study will also determine the independent effects of OSA and obesity on insulin resistance and blood vessel function.

DETAILED DESCRIPTION:
OSA is a common sleep disorder that is characterized by a brief collapse of the upper airway during sleep. This blockage prevents air from flowing properly into the lungs and causes pauses in breathing. If left untreated, OSA can cause high blood pressure, memory problems, weight gain, impotency, and headaches. It is also associated with an increased risk of inflammation-related heart conditions. Obesity is common among individuals with OSA and it may also be associated with inflammation. It is not known, however, whether the increased risk of heart problems is caused primarily by the inflammatory effects of OSA or obesity.

The most common treatment for OSA is continuous positive airway pressure (CPAP) therapy, in which a mask is worn over the nose during sleep. Air flows through the mask to maintain a level of pressure that keeps the throat open. The most common treatment for obesity is weight loss. This study will determine the primary cause of heart-related inflammation by evaluating the individual and combined effects of CPAP therapy and a weight loss program in treating obese individuals with OSA. The study will also determine the independent effects of these therapies on insulin resistance and blood vessel function (arterial stiffness, central arterial pressures).

This study will enroll obese individuals with moderate to severe OSA for a total of 24 weeks. Potential participants will first take part in an overnight sleep study at the University of Pennsylvania sleep lab. Sensors will monitor body functions during the night, including brain and muscle activity, eye movement, heart rate, breathing effort, air flow, and blood oxygen levels. Eligible participants will then be randomly assigned to CPAP therapy, a weight loss program, or a combination of the two. Participants in the weight loss program will receive weekly dietary counseling and will be encouraged to decrease caloric intake and increase physical activity. Participants receiving CPAP therapy will use a CPAP machine each night while they sleep. Study visits for all participants will occur at baseline and Weeks 6, 12, and 24. Blood will be collected to measure levels of triglycerides, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, and levels of C-reactive protein (CRP), which is an inflammation biomarker. Insulin resistance will be evaluated using a glucose tolerance test, and blood vessel function will be evaluated using a brachial artery reactivity test in which artery size and blood flow will be measured with an ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe OSA (as defined by an apnea-hypopnea index [AHI] score greater than 15 events per hour)
* Body mass index greater than 30 kg/m
* Baseline CRP greater than 1.0 mg/dL

Exclusion Criteria:

* Predominant central sleep apnea
* Type 1 Diabetes
* Type 2 Diabetes associated with either: (a) unstable anti-diabetic therapy (anti-diabetic medication changes within past 3 months); (b) Hemoglobin A1C levels > 7%; (c) Inability to perform home blood glucose monitoring (fingerstick checks).
* Requires use of supplemental oxygen
* Acute coronary syndrome or stroke in the 3 months prior to study entry
* A high-risk occupation or motor vehicle driving record, as defined by a score of 10 points or higher on an occupational and driving habits questionnaire
* Blood pressure greater than 160/95 mm Hg (may be re-screened after blood pressure control is obtained)
* Active infection, cancer, or chronic inflammatory disorder
* Use of systemic steroids
* Currently on an unstable dose of statin therapy (participants taking statins must be on a stable dose for at least 8 weeks prior to study entry)
* Simultaneous use of peroxisome proliferator-activated receptor (PPAR)-alpha (e.g., gemfibrozil, fenofibrate) or PPAR-gamma (e.g., rosiglitazone, pioglitazone)
* Consumes more than 14 alcoholic drinks per week
* History of surgery in the 3 months prior to study entry
* Sustained ventricular or supraventricular tachycardia greater than 30 seconds during overnight sleep study
* Known left ventricular ejection fraction less than 30% or decompensated congestive heart failure requiring hospitalization in the year prior to study entry
* Any episode of decompensated respiratory function requiring hospitalization in the year prior to study entry
* Severe restless leg syndrome or chronic pain syndrome that gives rise to frequent awakenings at night, as determined during the overnight sleep study (individuals may still be enrolled if these sleep-disrupting disorders can be resolved prior to study entry)
* Pregnant or likely to become pregnant (i.e., pre-menopausal and not using a form of birth control)
* Severe depression, as defined by a score of 29 or higher on the Beck Depression Index, or suicidal ideation
* Serious medical or psychological condition that may compromise the participant's safety or successful participation in the study, in the opinion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2006-09; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio A. Chirinos, MD, Principal Investigator — University of Pennsylvania, Philadelphia Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Jain S, Gurubhagavatula I, Townsend R, Kuna ST, Teff K, Wadden TA, Chittams J, Hanlon AL, Maislin G, Saif H, Broderick P, Ahmad Z, Pack AI, Chirinos JA. Effect of CPAP, Weight Loss, or CPAP Plus Weight Loss on Central Hemodynamics and Arterial Stiffness. Hypertension. 2017 Dec;70(6):1283-1290. doi: 10.1161/HYPERTENSIONAHA.117.09392. Epub 2017 Oct 16. PMID 29038203
- [Derived] Chirinos JA, Gurubhagavatula I, Teff K, Rader DJ, Wadden TA, Townsend R, Foster GD, Maislin G, Saif H, Broderick P, Chittams J, Hanlon AL, Pack AI. CPAP, weight loss, or both for obstructive sleep apnea. N Engl J Med. 2014 Jun 12;370(24):2265-75. doi: 10.1056/NEJMoa1306187. PMID 24918371

RESULTS

PARTICIPANT FLOW:
Groups:
- CPAP: Participants will receive CPAP therapy.
  CPAP therapy: Participants receiving CPAP therapy will use a CPAP machine each night while they sleep.
- Weight Loss: Participants will take part in a weight loss program.
  Weight Loss Program: Participants in the weight loss program will receive weekly dietary counseling and will be encouraged to decrease caloric intake and increase physical activity.
- Combination: Participants will receive CPAP therapy and take part in a weight loss program.
  Weight Loss Program: Participants in the weight loss program will receive weekly dietary counseling and will be encouraged to decrease caloric intake and increase physical activity.
  CPAP therapy: Participants receiving CPAP therapy will use a CPAP machine each night while they sleep.
Period: Overall Study
Arm/Group | CPAP | Weight Loss | Combination
Started | 58 | 61 | 62
Completed | 48 | 42 | 46
Not Completed | 10 | 19 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP | Weight Loss | Combination | Total
Number analyzed (Participants) | 58 | 61 | 62 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (10) | 48.3 (10) | 49 (10) | 49 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 29 | 77
  Male | 35 | 36 | 33 | 104
Region of Enrollment [Number; unit: participants]
  United States | 58 | 61 | 62 | 181

OUTCOME MEASURES:

1. Primary Outcome: Inflammation
Time Frame: Measured at Baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: percentage of change in crp at week 24
Groups:
- CPAP - Adherent: Participants will receive CPAP therapy.
  CPAP therapy: Participants receiving CPAP therapy will use a CPAP machine each night while they sleep.
- Weight Loss - Adherent: Participants will take part in a weight loss program.
  Weight Loss Program: Participants in the weight loss program will receive weekly dietary counseling and will be encouraged to decrease caloric intake and increase physical activity.
- Combination - Adherent: Participants will receive CPAP therapy and take part in a weight loss program.
  Weight Loss Program: Participants in the weight loss program will receive weekly dietary counseling and will be encouraged to decrease caloric intake and increase physical activity.
  CPAP therapy: Participants receiving CPAP therapy will use a CPAP machine each night while they sleep.
Arm/Group | CPAP - Adherent | Weight Loss - Adherent | Combination - Adherent
Number analyzed (Participants) | 48 | 42 | 46
percentage of change in crp at week 24 | -11.47 [-26.09 to 6.03] | -37.45 [-49.23 to -22.94] | -32.66 [-47.14 to -14.22]

2. Secondary Outcome: Change in Insulin Resistance (Insulin Sensitivity Index, x10-4/Min-1/μU/ml)
Description: Assessed using the frequently sampled intravenous glucose tolerance test (FSIGTT) which evaluates blood glucose and insulin levels. Insulin sensitivity is estimated using the Bergman's minimal model.
Time Frame: Measured at Baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: x10-4/min-1/μU/ml
Groups:
- Weight Loss - Adherent: Participants will receive take part in a weight loss program.
  Weight Loss Program: Participants in the weight loss program will receive weekly dietary counseling and will be encouraged to decrease caloric intake and increase physical activity.
Arm/Group | CPAP - Adherent | Weight Loss - Adherent | Combination - Adherent
Number analyzed (Participants) | 48 | 42 | 46
x10-4/min-1/μU/ml | .06 [-.34 to .46] | .43 [-.04 to .9] | .74 [.24 to 1.23]

3. Secondary Outcome: Change in LDL Cholesterol Levels
Time Frame: Measured at Baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | CPAP - Adherent | Weight Loss - Adherent | Combination - Adherent
Number analyzed (Participants) | 48 | 42 | 46
mg/dL | -3.76 [-10.08 to 2.55] | -9.25 [-16.87 to -1.6] | -13.54 [-22.03 to -5.05]

4. Secondary Outcome: Change in Triglyceride Levels
Time Frame: Measured at Baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | CPAP - Adherent | Weight Loss - Adherent | Combination - Adherent
Number analyzed (Participants) | 48 | 42 | 46
mg/dL | -7.1 [-24.2 to 10] | -23.2 [-43.8 to -2.6] | -53 [-76 to -30.2]

5. Secondary Outcome: Change in HDL Cholesterol Levels
Time Frame: Measured at Baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | CPAP - Adherent | Weight Loss - Adherent | Combination - Adherent
Number analyzed (Participants) | 48 | 42 | 46
mg/dL | -0.62 [-2.74 to 1.5] | 0.71 [-1.85 to 3.27] | 0.49 [-2.37 to 3.34]

ADVERSE EVENTS:
Description: Clustered data collection. Data on separate Adverse Event Terms not available. All adverse events were non serious so they are reported under Other Adverse Events.
Arm/Group | CPAP | Combination | Weight Loss
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 10/58 | 10/62 | 9/61
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CPAP (N=58) | Combination (N=62) | Weight Loss (N=61)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 — Nasal or sinus congestion
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 8
Flu (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nostril Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Worsening of Respiratory Allergy Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
"Shakiness" After IVGTT (Nervous system disorders) | 0 | 2 | 0
Burning Sensation after IVGTT (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lump at site of IV (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bruising/Tenderness- IV (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Vomited during IVGTT (Gastrointestinal disorders) | 0 | 0 | 1
Rash from Lead (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eye Irritation (Eye disorders) | 0 | 3 | 0
High Blood Pressure (Cardiac disorders) | 0 | 1 | 1
Chest Pain (Cardiac disorders) | 1 | 2 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngitis (Ear and labyrinth disorders) | 0 | 1 | 0
Type II Diabetes (Endocrine disorders) | 0 | 2 | 0
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 | 2 | 0
Self Committed to Hospital (General disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Tendonitis of Shoulder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling in legs and ankles (Cardiac disorders) | 1 | 0 | 0
Knee Replacement Surgery (Surgical and medical procedures) | 1 | 0 | 0
Wisdom Teeth Removal (Surgical and medical procedures) | 0 | 1 | 0
Rotator Cuff Surgery (Surgical and medical procedures) | 0 | 0 | 1
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Leg Cramps (Cardiac disorders) | 0 | 1 | 0
Panic Attack (Psychiatric disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pain in ankle/ lower back (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dehydration (General disorders) | 1 | 0 | 0
Sprained Wrist/ Bruised Knee (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Right Flank Pain (General disorders) | 0 | 1 | 0
Tooth Extraction and Implant (Surgical and medical procedures) | 1 | 0 | 0
Possible Urinary Tract Infection (Renal and urinary disorders) | 0 | 1 | 0
New diagnosis of fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intestinal Cramping (Gastrointestinal disorders) | 0 | 1 | 0
Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ankle Injury (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Abdominal Pain/ Kidney Stone (Renal and urinary disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No